CLINICAL TRIAL: NCT07362797
Title: Comparison of Clinical Application of Right Visual Double Lumen Tube and Right Ordinary Double Lumen Tube in Thoracoscopic Surgery for Adult Patients
Brief Title: Clinical Application of Right Visual Double Lumen Tube in Thoracoscopic Surgery for Adult Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diansan Su (Other)
Collaborators: Ningbo No.2 Hospital (Other); Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Sponsor-Investigator, Diansan Su, Chief Physician, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZJU2025C144
Record Dates: First submitted 2026-01-07; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Thoracoscopic Surgery; Double Lumen Tube Intubation
Keywords: double lumen tube; FOB; thoracoscopic surgery; Visual dual-lumen tube

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual double-lumen tube group (Active Comparator): Lung-isolation thoracoscopic surgery using a right-side visual double-lumen tube.
  Interventions: Device: visible double-lumen tube
- Non-visual dual-lumen tube (ordinary dual-lumen tube) group (Active Comparator): Lung isolation thoracoscopic surgery was performed with fiberoptic bronchoscopy assistance using a standard double-lumen tube on the right side (non-visual double-lumen tube).
  Interventions: Device: lumen intubation tube

INTERVENTIONS:
Device: visible double-lumen tube — A visible double-lumen tube on the right side
  Other Names: visible double-lumen tube group
  Arms: visual double-lumen tube group
Device: lumen intubation tube — The standard double-lumen tube on the right side was positioned with the aid of a fiberoptic bronchoscope.
  Other Names: lumen intubation tube group
  Arms: Non-visual dual-lumen tube (ordinary dual-lumen tube) group

SUMMARY:
This clinical trial aims to understand whether a visual double-lumen intubation tube can improve the first-attempt success rate and reduce complications compared to a standard double-lumen tube. The trial primarily aims to answer the following questions:

Does a double-lumen tube improve the first-attempt success rate?

Does a visual double-lumen tube reduce the likelihood of obstruction of the right upper lobe bronchial opening?

Does a visual double-lumen tube require fewer adjustments during surgery?

Do patients with visual double-lumen tubes experience fewer perioperative complications compared to those with standard double-lumen tubes?

Participants will:

Use a visual double-lumen tube partially and a standard double-lumen tube partially.

Record the perioperative status of all patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: at least 18 years old, gender is not limited.
* American Anesthesiologists Association (ASA) Grade I-III;
* Elective Video-Assisted Thoracoscopic Lobectomy.
* Informed consent of the patient or family member.
* People who are willing to accept perioperative visits.

Exclusion Criteria:

* Patients with contraindications for right double-lumen tube insertion (such as right bronchial tumor).
* The patient has known tracheobronchial anatomical abnormalities
* Patients previously diagnosed or suspected of having airway difficulty.
* Patients who need rapid sequence induction.
* Patients requiring emergency surgery
* Patients who have undergone thoracic surgery, systemic infection or suspected tuberculosis in the past four weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary purpose | After anesthesia induction, the laryngoscope is inserted and the timing begins until the endotracheal tube position is confirmed. The endotracheal tube is then fixed, and mechanical ventilation is initiated (approximately 10 minutes).
  To study whether the right visual double lumen tube can improve the success rate of initial intubation compared with the right ordinary double lumen tube.

SECONDARY OUTCOMES:
Secondary purposes | After the endotracheal tube is secured, the patient is ventilated by a ventilator, and ventilation of the right single lung is initiated (lasting approximately 2-3 minutes).
  Compare the obstruction of the right upper bronchial opening in the two groups of patients.
Intraoperative cannulation position adjustment | The entire surgery (approximately 1-3 hours).
  Compare the number of times the endotracheal intubation position needed to be adjusted and the total adjustment time between the two groups of patients.
postoperative complications | From the end of surgery to the patient's discharge (2-3 days).
  The postoperative complications of the two groups of patients were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine,, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided